CLINICAL TRIAL: NCT00360269
Title: Atomoxetine Treatment for ADHD and Marijuana Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Aimee McRae-Clark, Associate Professor of Psychiatry, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21DA018221 (NIH); R21DA018221 (NIH); NCT00227851 (obsolete NCT alias)
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Marijuana Abuse; Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Marijuana Abuse; Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Motivational Interviewing; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Atomoxetine plus Motivational Enhancement Therapy
  Interventions: Drug: Atomoxetine; Procedure: Motivational enhancement therapy
- Placebo (Placebo Comparator): Placebo plus Motivational Enhancement Therapy
  Interventions: Procedure: Motivational enhancement therapy; Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — 25 to 100 mg daily
  Other Names: Strattera
  Arms: Active
Procedure: Motivational enhancement therapy — Three sessions
  Other Names: MET
Drug: Placebo — 25 to 100 mg daily
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The aim of the study is to determine if atomoxetine treatment combined with motivational enhancement therapy is effective in reducing marijuana use in adult individuals with attention-deficit hyperactivity disorder and marijuana dependence.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the medication atomoxetine, or Strattera, plus 3 sessions of counseling can help people to reduce the symptoms of ADHD and to help cut back on their marijuana use. Participation in the study is approximately 12 weeks of medication treatment and doctor's visits once a week. The first 2 visits consist of evaluations to determine if you qualify to participate. These visits are approximately 2-3 hours long and will include questions about your past and present substance use, psychiatric history, a routine physical exam, bloodwork, and paper and pencil questionnaires about your marijuana use. Once you are enrolled in the study, visits are typically 30 minutes long, once a week. The one-on-one counseling sessions regarding marijuana use are 1 hour long and you will have 3 sessions throughout the study. If you qualify for this study, you will receive either atomoxetine, or a placebo (sugar pill). Study participants will have a 50% chance of receiving atomoxetine. Atomoxetine is a non-stimulant, commonly used to treat ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women, 18 to 65 years of age
2. Meet DSM-IV criteria for marijuana dependence
3. Meet DSM-IV criteria for current ADHD, determined by a clinical interview and confirmed by semi-structured interview with the Conners' Adult ADHD Diagnostic Interview for DSM-IV (CAAR-D; Conners et al, 1999)
4. ADHD symptom severity indicated by a score of 12 or greater on the Wender-Reimherr Adult Attention Deficit Disorder Scale
5. ADHD symptoms must be corroborated by a second informant on either current symptoms (by a significant other or close friend) or childhood symptoms (by a parent or older sibling)
6. All subjects will agree to and sign a written, IRB-approved informed consent
7. Subjects must live within a 60-mile radius of Charleston, SC, to facilitate study visit compliance

Exclusion Criteria:

1. Individuals meeting DSM-IV dependence for a substance other than marijuana with the exception of nicotine and caffeine. Dependence on nicotine and caffeine will be allowed since dependence on these substances commonly co-occurs with marijuana dependence and excluding these individuals would compromise study recruitment
2. Individuals meeting DSM-IV criteria for a lifetime history of schizophrenia or another non-affective psychotic disorder or bipolar disorder, since these patients will most likely be taking other psychotropic medications and often require intensive psychiatric care
3. Individuals meeting DSM-IV criteria for current major depressive disorder or eating disorder, since these individuals will likely require treatment with psychotropic medications. Subjects may meet criteria for a minor mood disorder (dysthymia) and for anxiety disorders. The inclusion of subjects with these disorders will be allowed as they commonly co-exist among patients with marijuana dependence (Stephens et al, 1993)
4. Individuals who present significant suicidal risk
5. Individuals with significant cognitive impairment as measured by a score of less than 26 on the Mini-Mental Status Exam, as they may be unable to understand the informed consent, comply with study protocol, or accurately complete assessments
6. Individuals currently receiving stimulants, benzodiazepines, antidepressant or antipsychotic medications, as these medications could confound the effects of atomoxetine treatment
7. Individuals currently receiving psychotherapy focusing on reducing marijuana use or on ADHD symptoms, as this could confound the effects of atomoxetine treatment. Participation in 12-step programs will be allowed
8. Pregnant or nursing women, or women who refuse to use adequate birth control, as atomoxetine has not been approved for use in pregnancy
9. Individuals without stable housing, as contacting these individuals would be difficult
10. Individuals with major medical illnesses (e.g., HIV, renal failure, unstable angina, chronic obstructive pulmonary disease, infectious hepatitis)
11. Patients with hypertension (defined as having blood pressure greater than 140/90 measured on 3 or more occasions), as atomoxetine treatment can be associated with increases in blood pressure
12. Patients with evidence of hepatic insufficiency, as atomoxetine requires hepatic metabolism
13. Patients with urinary hesitancy or urinary hesitation, as atomoxetine has been associated with some urinary hesitation in clinical trials
14. Individuals who, in the investigators' opinion, would not be able to comply with study procedures, such as individuals unable to reliably present for intake appointments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee L McRae, PharmD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Chauchard E, Hartwell KJ, McRae-Clark AL, Sherman BJ, Gorelick DA. Cannabis Withdrawal in Adults With Attention-Deficit/Hyperactivity Disorder. Prim Care Companion CNS Disord. 2018 Feb 22;20(1):17m02203. doi: 10.4088/PCC.17m02203. PMID 29489073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited between November 2005 and June 2008 primarily through media advertisements and fliers
Groups:
- Atomoxetine; Placebo: Flexible dose up to 100mg/day
Period: Overall Study
Arm/Group | Atomoxetine | Placebo
Started | 19 | 19
Completed | 9 | 7
Not Completed | 10 | 12
Not completed — Lost to Follow-up | 7 | 9
Not completed — Physician Decision | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (10.0) | 30.4 (13.0) | 29.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 16 | 13 | 29
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Secondary Outcome: Self-reported Longitudinal Use
Description: Participants' self-report of mean frequency of use of marijuana from baseline through week 12 visit of the study was assessed using a Time-Line Follow-Back.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage of days used
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 19 | 19
Percentage of days used | 60.1 (31.5) | 68.1 (31.3)

2. Primary Outcome: Estimated Week 12 Self-reported Use
Description: Participants' self-report of mean frequency of use of marijuana during week 12 of the study was assessed using a Time-Line Follow-Back.
Time Frame: One week (study week 12)
Measure: Mean (Standard Error); unit: Times per day
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 19 | 19
Times per day | 2.17 (.34) | 1.84 (.34)

3. Secondary Outcome: Urine Drug Screens
Description: Participants submitted a urine sample weekly. Percentage of marijuana positive urine samples were calculated per group.
Time Frame: 12 weeks
Measure: Number; unit: Percentage of positive UDS
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 19 | 19
Percentage of positive UDS | 87.3 | 85.3

4. Secondary Outcome: Wender-Reimherr Adult Attention Deficit Disorder Scale
Description: The WRAADDS is intended to measure the severity of ADHD symptoms in adults. It measures symptoms in seven categories: attention difficulties, hyperactivity/restlessness, temper, affective lability, emotional over-reactivity, disorganization, and impulsivity. The scale rates individual items from 0-2 (0=not present, 1=mild, 2=clearly present), with a minimum score of 0 and maximum score of 46. Reported here is change from Baseline to Week 12 (or LOCF).
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 19 | 19
Units on a scale | -15.05 (10.96) | -11.05 (7.59)

5. Secondary Outcome: Clinical Global Impression, Improvement Scale
Description: The Clinical Global Impression - Improvement scale (CGI-I) was used to assess improvement in ADHD symptoms during study participation. CGI-I is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 19 | 19
Units on a scale | 2.63 (0.68) | 3.26 (0.93)

ADVERSE EVENTS:
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 19/19 | 16/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atomoxetine (N=19) | Placebo (N=19)
Anxiety/depression (Psychiatric disorders) | 3 | 2
Dizziness/lightheaded (Nervous system disorders) | 6 | 3
Drowsiness (Nervous system disorders) | 3 | 3
Dry mouth (General disorders) | 3 | 3
Gastrointestinal (Gastrointestinal disorders) | 9 | 4
Headache (Nervous system disorders) | 7 | 5
Hot/cold flashes (General disorders) | 3 | 0
Increased urination (Renal and urinary disorders) | 0 | 2
Insomnia (General disorders) | 0 | 4
Irritability (Psychiatric disorders) | 2 | 1
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 6 | 5
Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sexual dysfunction (Reproductive system and breast disorders) | 5 | 0
Sinus/allergies/flu-like symptoms (General disorders) | 7 | 9
Other (General disorders) | 5 | 3

LIMITATIONS AND CAVEATS:
Small sample size and poor retention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No